CLINICAL TRIAL: NCT01588977
Title: Subchondral Microfracture of Tibia After Arthroscopic Anterior Cruciate Ligament Surgery Reconstruction With Two Different Drilling Techniques. Correlation With Postoperative Pain
Brief Title: Subchondral Microfracture of Tibia After Arthroscopic Anterior Cruciate Ligament Surgery Reconstruction
Status: Completed | Type: Observational
Sponsor: Hospital Ambroise Paré Paris (Other)
Responsible Party: Principal Investigator, Shahnaz Klouche, MD, Physician Clinical Research, Hospital Ambroise Paré Paris
Other Study IDs: APR042012
Record Dates: First submitted 2012-04-27; First posted 2012-05-01 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Anterior Cruciate Ligament Reconstruction; Subchondral Microfractures of Tibia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- All-Inside TightRope technique
- ACL reconstruction with TLS system
- Hamstring Tendon Graft Reconstruction of the ACL

SUMMARY:
The arthroscopic anterior cruciate (ACL) ligament reconstruction surgery is widespread. The creation of the tibial tunnel, retrograde or antegrade, is not consensual. A cadaveric study demonstrated tibial subchondral microfractures in the group "antegrade tibial tunnel" unlike group "retrograde tibial tunnel." To our knowledge, no clinical evaluation was performed. The investigators hypothesize that retrograde drilling will cause less local bone injury than antegrade drilling in creation of the tibial tunnel for ACL reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* arthroscopic reconstruction surgery of an Anterior Cruciate Ligament tear

Exclusion Criteria:

* previous reconstruction of ACL
* associated lesions (meniscal tear, other ligament...)
* Refusal consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary arthroscopic reconstruction surgery of an Anterior Cruciate Ligament tear
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2012-04; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Subchondral microfracture of tibia on MRI | 2 days after surgery

SECONDARY OUTCOMES:
Pain on Visual Analogue Scale | During two days after surgery, twice a day

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Ambroise Paré Hospital, Boulogne-Billancourt
  - Hôtel-Dieu CHU Nantes, Nantes
  - Polyclinique de L'Europe, Saint-Nazaire